CLINICAL TRIAL: NCT02102594
Title: Therapy of Antibody-mediated Autoimmune Diseases by Bortezomib (TAVAB)
Acronym: TAVAB
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: recruitment difficulties
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Prof. Dr. med. Falk Hiepe (Charité, Internal Medicine / Rheumathology) (Unknown); NeuroCure Clinical Research Center, Charite, Berlin (Other)
Responsible Party: Principal Investigator, Andreas Meisel, Prof. Dr., Charite University, Berlin, Germany
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TAVAB; 2013-005362-19 (EudraCT Number)
Record Dates: First submitted 2014-03-25; First posted 2014-04-03 (Estimated); Last update posted 2019-12-03 (Actual); Status verified 2019-11

CONDITIONS: Myasthenia Gravis; Systemic Lupus Erythematosus; Rheumatoid Arthritis
Keywords: Myasthenia Gravis; Systemic Lupus Erythematosus; Rheumatoid Arthritis; proteasome inhibitor; Bortezomib; Velcade; antibody-mediated autoimmune disease
MeSH Terms: conditions — Myasthenia Gravis; Lupus Erythematosus, Systemic; Arthritis, Rheumatoid | interventions — Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bortezomib (Velcade) (Experimental)
  Interventions: Drug: Bortezomib

INTERVENTIONS:
Drug: Bortezomib — Bortezomib will be subcutaneously applicated in 2 treatment cycles with 4 injections of 1.3 mg Bortezomib /m2 body surface per cycle.
  Other Names: Velcade

SUMMARY:
The aim of this pilot study is to investigate the application of proteasome inhibitor Bortezomib (Velcade®, approved for therapy of multiple myeloma) in patients with therapy-refractory antibody-mediated autoimmune diseases. The investigators hypothesis is that the proteasome inhibition will lead to reduced antibody titers and improved clinical outcome.

ELIGIBILITY:
(main) Inclusion Criteria:

* age 18 - 75 years at screening
* ability to give written consent, informed written consent
* negative pregnancy test at screening
* therapy-refractory Myasthenia Gravis (generalized) or Systemic Lupus Erythematosus or Rheumatoid Arthritis

(main) Exclusion Criteria:

* Belimumab therapy within the last 6 months
* B-cell-depletion therapy within the last 9 months
* heart or kidney insufficiency
* known intolerability to Bortezomib
* participation in another interventional trial within the last 3 months
* liver cirrhosis
* preexistent sensory or motor polyneuropathy ≥ degree 2 (NCI CTC AE criteria), within 14 days before screening
* hints on clinically apparent herpes zoster reactivation
* active systemic infection, or viral infection (CMV, EBV) within last 6 month before screening
* serologically active hepatitis B and /or C, known HIV infection
* tumor disease currently or within last 5 years
* clinically relevant liver, kidney or bone marrow function disorder
* pregnancy or lactation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2014-10; Primary Completion 2019-08-30 (Actual); Study Completion 2019-08-30 (Actual)

PRIMARY OUTCOMES:
change in disease specific antibody titers after application of Bortezomib | 6 months after end of therapy (6 weeks) compared to baseline (before therapy)
  Change in disease specific antibody titers (anti-ACh for myasthenia gravis, anti-dsDNA for systemic lupus erythematosus, anti-ACPA for rheumatoid arthritis) 6 months after end of Bortezomib therapy (duration 6 weeks) compared to baseline (before therapy).

SECONDARY OUTCOMES:
Change in disease specific antibody titer after Bortezomib application | at regular intervals up to 30 weeks compared to baseline
  Change in disease specific antibody titer after Bortezomib application (except at time point 6 months after end of therapy = primary outcome measure)
Change in quality of life (Qol score) | at regular intervals up to 30 weeks compared to baseline
Change in Activities of Daily Living (Adl score) | at regular intervals up to 30 weeks compared to baseline
change in dose of immunosuppressive co-medication | at regular intervals up to 30 weeks compared to baseline
Change in titers of protective antibodies (e.g. measles) | at regular intervals up to 30 weeks compared to baseline
  Change in titers of protective antibodies against measles virus, rubella virus, varicella zoster virus, pneumococcus, cytomegalovirus
Change in number of antibody producing plasmablasts/cells | at regular intervals up to 30 weeks compared to baseline
  Change in number of antibody producing plasmablasts/cells in peripheral blood
Change in concentration of soluble mediators (e.g. IL-6) | at regular intervals up to 30 weeks compared to baseline
  Change in concentration of soluble mediators (e.g. IL-6) in peripheral blood
need for hospitalisation | at regular intervals up to 30 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Meisel, Prof. Dr., Principal Investigator — Charité - Universitätsmedizin Berlin, NeuroCure Clinical Research Center; Falk Hiepe, Prof. Dr., Principal Investigator — Charité - Universitätsmedizin Berlin, Internal Medicine / Rheumatology
Locations (2):
- Germany (2):
  - Charite - Universitätsmedizin Berlin, NeuroCure Clinical Research Center, Berlin
  - Charité - Universitätsmedizin Berlin, Internal Medicine / Rheumathology, Berlin

REFERENCES:
- [Background] Kohler S, Losen M, Alexander T, Hiepe F, Meisel A. Myasthenia gravis: subgroup classifications. Lancet Neurol. 2016 Apr;15(4):356-7. doi: 10.1016/S1474-4422(16)00033-8. No abstract available. PMID 26971655
- [Background] Kohler S, Marschenz S, Grittner U, Alexander T, Hiepe F, Meisel A. Bortezomib in antibody-mediated autoimmune diseases (TAVAB): study protocol for a unicentric, non-randomised, non-placebo controlled trial. BMJ Open. 2019 Jan 28;9(1):e024523. doi: 10.1136/bmjopen-2018-024523. PMID 30696682